CLINICAL TRIAL: NCT07325721
Title: Hypofractionated Radiotherapy With a Focal Microboost for High-Risk and Locally Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104214; Pro00147655 (Other: MUSC IRB)
Record Dates: First submitted 2025-11-24; First posted 2026-01-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer; Prostate Cancer Patients Treated by Radiotherapy
Keywords: Prostate cancer; Microboost; hypofractionated
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hypofractationed pelvic radiation with microboost (Experimental)
  Interventions: Radiation: Hypofractionated radiation with a microboost

INTERVENTIONS:
Radiation: Hypofractionated radiation with a microboost — Patients will receive 25 fractions of external beam radiation therapy. Dose to the elective lymph nodes will be 45 Gy in 25 fractions. Dose to the prostate and portions of the seminal vesicles will be 68 Gy in 25 fractions. A microboost to up to three dominant intraprostatic nodules will be given in 25 fractions (dose range 70-83 Gy). Simultaneous integrated boost to sites of pelvic lymphadenopathy may be given. Androgen deprivation therapy will be per local standard of care.

SUMMARY:
This study is for adult men with previously untreated high risk, very high risk, or pelvic lymph node positive prostate cancer. The purpose of this study is to evaluate the safety and effectiveness of the combination of two emerging radiation treatment techniques (hypofractionated radiotherapy and microboost technique). Participation will include standard of care visits along with questionnaires and blood draws completed for research purposes. There is optional banking of blood and prostate biopsy tissue which will not require extra biopsies. Participation in this study is anticipated to last approximately 6 weeks with follow up every three months for two years then twice yearly for years 3-5.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Biologically male patients aged 18 years and older.
4. Ability to receive pelvic radiotherapy and be willing to adhere to the protocol regimen.
5. Previously untreated prostate cancer (with cytotoxic chemotherapy, cryotherapy, ablative treatment, surgical or radiation therapy). Prior transurethral resection of prostate (TURP) is permitted if 90 days or more prior to the start of radiotherapy.
6. Localized or locally advanced prostate cancer meeting NCCN criteria for high risk, very high risk or non-metastatic, pelvic lymph node positive defined as having at least one or more of the following:

   1. PSA >20 ng/mL prior to starting ADT.
   2. cT3a-T4 by digital exam or imaging.
   3. Gleason score of 8-10 (grade group 4 or 5).
   4. Staged as N1M0 by the treating investigator (pelvic lymph node positive, below the aortic bifurcation) based on soft tissue imaging within 120 days prior to registration (may include CT, MRI or PSMA PET/CT, of fluciclovine choline PET/CT).
7. History and physical exam within 120 days prior to registration.
8. ECOG performance status 0-2.
9. Be able to undergo MRI of the prostate and/or pelvis as a component of RT planning.
10. Have at least one MRI visible target for microboost (PI-RADS≥ 4 version 2.0).
11. Bone and soft tissue imaging as clinically indicated for staging within 120 days prior to registration.
12. For males: use of condoms or other methods to ensure effective contraception with partner during radiation and for six months after completion of radiation.
13. Adequate hematologic function within 120 days prior to registration as defined by:

    1. hemoglobin >=9.0 g/dL independent of transfusion, and
    2. platelet count >= 100,000 x 10 ^9/microliter independent of transfusion.
14. Adequate hepatic function within 120 days prior to registration defined as total bilirubin <2 x institutional upper limits of normal (ULN is 1.2 mg/dL). If labs are done at outside institution, total bilirubin should be <2.4.
15. Agreeable and eligible to receive long term (defined as 12-36 months) ADT as a standard component of prostate cancer therapy.

Exclusion Criteria:

* 1. Concurrent use of testosterone supplementation unless discontinued by time of registration.

  2. Definitive radiologic evidence of metastatic disease outside of the pelvic nodes on conventional imaging (bone scan, CT scan, MRI).

  3. Prior pelvic radiotherapy. 4. Pre-existing conditions or overall health status which disqualifies the patient from curative intent-RT. Patients with life expectancy less than 5 years are not eligible.

  5. Treatment with another investigational prostate cancer therapy within 12 months.

  6. Prior total prostatectomy, cryotherapy, high-intensity focused ultrasound, irreversible electroporation, MRI ablation, laser ablation, transurethral ultrasound ablation, aquablation directed towards the prostate for any prostate disease or condition.

  7. Prior or concurrent invasive pelvic malignancy (except non-melanomatous skin cancer) or lymphomatous or hematogenous malignancy, unless disease free for a minimum of 5 years.

  8. Any condition that, in the opinion of the investigator, would preclude participation in this study.

  9. Prior pharmacologic androgen ablation for prostate cancer is allowed only if the onset of androgen ablation (both LHRH agonist and oral anti-androgen) is ≤ 90 days prior to registration.

  10. Inability to undergo implantation of gold fiducial markers or rectal spacer gel.

  11. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2034-01-01 (Estimated)

PRIMARY OUTCOMES:
CTCAE grade 2 or higher acute genitourinary toxicity | 1 month post radiation

SECONDARY OUTCOMES:
grade 2 or higher acute GI toxicity, late GU toxicity and late GI toxicity | 5 years
PSA failure rate | 2 years
death from any cause | 5 years
Mean change in Sexual Health Inventory for Men (SHIM) score | 5 years
Mean change in EPIC-26 sexual domain score from baseline | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No